CLINICAL TRIAL: NCT01400009
Title: Vitamin D Replacement in Statin-Induced Myopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Mark Sherman, Associate Professor (Clinical), Dept of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-STAT-2010
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: HMG COA Reductase Inhibitor Adverse Reaction
Keywords: Statin; HMG COA Reductase Inhibitor; myalgia; vitamin D
MeSH Terms: conditions — Myalgia | interventions — Cholecalciferol; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects in this group will receive a placebo tablet (Lactose 100 mg) for the duration of the study
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): Subjects in this arm will receive a dose of 50,000 IU of vitamin D3, followed by weekly doses of 10,000 IU of vitamin D3
  Interventions: Drug: Vitamin D (Cholecalciferol )

INTERVENTIONS:
Drug: Vitamin D (Cholecalciferol ) — 10,000 IU tablets. 50,000 initial dose, followed by weekly doses of 10,000 IU
  Other Names: DIN number 00821772
  Arms: Vitamin D
Drug: Placebo — Standard Placebo made of Lactose 100 mg
  Other Names: Lactose 100 mg DIN 00501190
  Arms: Placebo

SUMMARY:
Pretreating people with replacement doses of vitamin D will allow them to tolerate Statin medications that have caused muscle pain for them in the past.

DETAILED DESCRIPTION:
Patients who have been unable to tolerate statin medications due to muscle pain will be randomly assigned to receive vitamin D or placebo for 6 weeks before reintroducing their statin medication. The investigators will judge whether vitamin D in the manner administered in the study reduces the myalgia with statins and allows patients to remain on these important medications.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults
* identified by their physician as having myalgia with their statin medication.

Exclusion Criteria:

* Unexplained CK > 4X upper limit of normal, at study entry, or on a statin medication in the past.
* Severe myositis
* Consumption in excess of 14 alcoholic beverages per week
* Situations which will cause difficulty in interpreting the vitamin D and / or PTH.

examples:

* Present consumption of vitamin D supplements > 1000 iu daily
* Renal impairment (Estimated creatinine clearance < 70 ± 14 mL/min/m2 in Males; and < 60 ± 10 mL/min/m2 in Females)
* Chronic liver disease or impaired liver function
* Any contraindication for statin re-challenge Example: rhabdomyolysis or allergy to statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
lack of need to stop statin medication due to myalgia | 12 weeks
  Ability to tolerate a statin at the same dosage that previously caused the individuals to stop due to myalgia

SECONDARY OUTCOMES:
reduction of visual analog pain score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Sherman, MD,CM, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC-Royal Victoria Hospital, Montreal, Quebec, Canada